CLINICAL TRIAL: NCT06542575
Title: Efficacy of the Integration of Digital Therapeutics and Home-based Cardiac Rehabilitation in High-Risk Post-PCI Patients on Cardiovascular Health
Brief Title: Efficacy of the Integration of Digital Therapeutics and Home-based Cardiac Rehabilitation in High-Risk Post-PCI Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yong He, Professor, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WestChinaH-CVD-006
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DTx-guided HBCR group (Experimental)
  Interventions: Other: DTx-guided HBCR
- Usual care group (No Intervention)

INTERVENTIONS:
Other: DTx-guided HBCR — The Huaxiaoxin WeChat mini program incorporating the core components of guidelines are divided into two main sections. Section 1 comprises interventions such as exercise training, educational programmes and cardiovascular risk factor management. Section 2 provides a secure platform for individualized feedback, just-in-time two-way communication, remote data transmission, and data repository, allowing patients and healthcare providers to access all relevant files anytime and anywhere throughout the 12-month study period.
  Arms: DTx-guided HBCR group

SUMMARY:
The DTx-HBCR trial will randomize 366 high-risk patients who undergo PCI at the West China Hospital of Sichuan University to either the 6-month DTx-guided HBCR group (intervention group) or the 6-months usual care group (control group) in a parallel-arm randomized controlled trial. The primary outcome is the difference between the intervention group and control group in walk distance on the 6-minute walk test (i.e., functional capacity) at 6 months post randomization. The key secondary outcomes include improvements in cardiovascular risk factor control, quality of life, psychological status, physical activity, major adverse cardiovascular events, and medication adherence. This study aims to evaluate the DTx-guided HBCR, a software-driven, multidisciplinary health intervention as an alternative to traditional in-center CR in patients with high-risk patients following percutaneous coronary intervention (PCI) compared with usual care alone.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, a participant must meet all of the following criteria:

  1. Women or men, the ages of 18 and 75 years.
  2. Have sufficient reading and writing language skills in Chinese.
  3. Be willing to participate the study and sign informed consent.
  4. Patients must have at least one clinical feature and one angiographic feature:

A. Clinical features: age ≥ 65 years, female sex, troponin positive acute coronary syndrome, established vascular disease (prior myocardial infarction, coronary revascularization or peripheral arterial disease) , diabetes mellitus requiring medication and chronic kidney disease (estimated glomerular filtration rate < 60 ml/min/1.73 m2 or creatinine clearance < 60 cc/min) .

B. Angiographic features: multivessel coronary artery disease, total stent length > 30 mm, thrombotic target lesion, bifurcation lesion requiring two stents, obstructive left main or proximal left anterior descending lesion and calcified target lesion requiring atherectomy.

Exclusion Criteria:

* A potential participant who meets any of the following criteria will be excluded from participation in this study:

  1. Contraindications to exercise rehabilitation (e.g., untreated ventricular tachycardia, severe heart failure (New York Heart Association class III or IV heart failure, or ejection fraction < 40%), uncontrolled hypertension or hypotension, active hemorrhage, severe liver failure, significant exercise limitations).
  2. Vision, hearing, cognition-related or mental impairment leading to inability to cooperate.
  3. Patients with established planned Phase II PCI.
  4. Having pre-existing comorbid disease with a life expectancy of < 1 year.
  5. Poor compliance and unable to complete the expected follow-up.
  6. Unable to access WeChat via a smartphone after training.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walk distance (i.e., functional capacity) at 6 months post randomization | At 6 months post randomization
  Change in distance participants walked (i.e., functional capacity) between the intervention and usual care groups, as measured by the 6MWT at 6 months postrandomization.

SECONDARY OUTCOMES:
Change in functional capacity at 3 months postrandomization | At 3 months postrandomization
  Change in distance participants walked (i.e., functional capacity) between the intervention and usual care groups, as measured by the 6MWT at 3 months postrandomization.
Change in conventional CVD risk factors at 3, 6 months post randomization | At 3, 6 months post randomization
  Changes in conventional CVD risk factors, such as lipid profile, glycosylated hemoglobin, BMI, BP, and smoking habits.
Change in quality of life at 3, 6 months post randomization | At 3, 6 months post randomization
  Quality of life as assessed by the Seattle Angina Questionnaire41 and the EuroQol 5-Dimensions Questionnaire.
Change in psychological status at 3, 6 months post randomization | At 3, 6 months post randomization
  Depression scores, as assessed by the 9-item Patient Health Questionnaire; anxiety scores, as assessed by the 7-item Generalized Anxiety Disorder questionnaire.
Change in physical activity levels at 3, 6 months post randomization | At 3, 6 months post randomization
  Qhysical activity levels as assessed by the International Physical Activity Questionnaire.
Change in medication adherence at 3, 6 months post randomization | At 3, 6 months post randomization
  Medication adherence as assessed by the 8-item Morisky Medication Adherence Scale.

OTHER OUTCOMES:
The incidence of major adverse cardiovascular events (MACEs) at 1 year post randomization | At 1 year post randomization
  MACEs, defined as the composite of cardiac death (namely, all deaths with a clear cardiovascular or unknown cause will be classified as cardiac, non-cardiac deaths is only due to a documented non-cardiac cause (e.g., cancer)), nonfatal myocardial infarction, nonfatal stroke, and target vessel revascularization.
User satisfaction | At 6 months post randomization
  User satisfaction as assessed the System Usability Scale modified for the Huaxiaoxin program.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF, CSR

REFERENCES:
- [Derived] Ma S, Chen Z, Zhang J, Liu J, Xu L, Huang B, Zhou M, Wang H, Chen Y, Wang M, Li C, He Y; DTx-HBCR trial investigators. Evaluation of the efficacy of integrating digital therapeutics with home-based cardiac rehabilitation on cardiovascular health in high-risk post-PCI patients (DTx-HBCR): Study protocol for a randomized controlled trial. Digit Health. 2025 Jul 25;11:20552076251360885. doi: 10.1177/20552076251360885. eCollection 2025 Jan-Dec. PMID 40735550